CLINICAL TRIAL: NCT01569594
Title: CorMatrix® ECM® for Carotid Repair Following Endarterectomy Registry
Brief Title: CorMatrix ECM for Carotid Repair Following Endarterectomy Registry
Status: Completed | Type: Observational
Sponsor: Elutia Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 11-PR-1021
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Carotid Stenosis
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Carotid Endarterectomy Subjects: Subjects undergoing patch angioplasty of the carotid artery following carotid endarterectomy using the CorMatrix ECM for Carotid Repair
  Interventions: Device: CorMatrix ECM for Carotid Repair

INTERVENTIONS:
Device: CorMatrix ECM for Carotid Repair — Subjects must be undergoing carotid endarterectomy with patch angioplasty closure

SUMMARY:
Assess device performance data from subjects undergoing patch angioplasty of the carotid artery following carotid endarterectomy using the CorMatrix ECM for Carotid Repair.

DETAILED DESCRIPTION:
The objective of this registry is to capture and assess device performance data from subjects undergoing patch angioplasty of the carotid artery following carotid endarterectomy using the CorMatrix ECM for Carotid Repair per its FDA cleared Indications for Use. This registry provides an ongoing post-market surveillance mechanism to document clinical outcomes on the use of the CorMatrix ECM for Carotid Repair.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be undergoing carotid endarterectomy with patch angioplasty closure.
* Subject's operative surgeon intends to use CorMatrix ECM as the patch material for closure of the carotid artery per its FDA cleared Indications for Use.
* The subject must possess the ability to provide written Informed Consent.
* The subject must express an understanding and willingness to fulfill all of the expected requirements of this clinical protocol.

Exclusion Criteria:

* Subjects with a known sensitivity to porcine material.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 230 subjects may be enrolled from up to ten U.S. clinical sites
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2012-04; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Cardio-Thoracic Surgeons, P.C. Trinity, Birmingham, Alabama
  - Vascular Surgical Associates P.C., Marietta, Georgia
  - Cardiac Surgery Associates, Indianapolis, Indiana
  - St Luke's Hospital, Kansas City, Missouri
  - Cardiovascular Surgery Clinic, PLLC, Memphis, Tennessee
  - UVA Heart and Vascular Center, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Subjects undergoing carotid endarterectomy with patch angioplasty closure using the CorMatrix ECM as the patch material.
Period: Overall Study
Arm/Group | Single Arm
Started | 230
Completed | 163
Not Completed | 67
Not completed — Physician Decision | 4
Not completed — Death | 13
Not completed — Lost to Follow-up | 22
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 13
Not completed — Other | 4
Not completed — No ECM used | 9

BASELINE CHARACTERISTICS:
Arm/Group | Carotid Endarterectomy Subjects
Number analyzed (Participants) | 221
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 221
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 203
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 221
Co-Morbidity Risk Factors [Count of Participants; unit: Participants]
  Hypertension | 182
  COPD | 32
  Diabetes | 84
  Chronic Renal Failure | 19
  CHF | 19
  Valve Disease | 9
  Previous AF | 22
  Previous MI | 45
  Previous TIA | 51
  Previous TIA - Symptomatic | 22
  Previous Stroke | 43
  Previous Stroke - Symptomatic | 20
  Obesity | 47
  Smoking | 75
  Previous Neck Surgery | 34
  Previous Neck Radiation | 2

OUTCOME MEASURES:

1. Primary Outcome: Carotid Procedure and Device Related Adverse Events to Determine Device Performance
Time Frame: 2 years
Measure: Number; unit: Device related adverse events
Arm/Group | Carotid Endarterectomy Subjects
Number analyzed (Participants) | 221
Device related adverse events
  Not related to device | 53
  Possibly related to device | 10
  Probably related to device | 1
  Definitely related to device | 2

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 13/221
Serious Adverse Events (participants affected / at risk) | 25/221
Other Adverse Events (participants affected / at risk) | 0/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=221)
GI bleed (Gastrointestinal disorders) | 1 (1)
Hematoma (Blood and lymphatic system disorders) | 4 (4)
CVA (Cardiac disorders) | 5 (5)
Blown carotid patch (Product Issues) | 1 (1)
Orthostatic hypotension episodes (Cardiac disorders) | 1 (1)
Post-op hoarseness from intubation (Surgical and medical procedures) | 1 (1)
Migraine (General disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Herald Bleed (Product Issues) | 1 (1)
VATS (Surgical and medical procedures) | 1 (1)
Restenosis (Cardiac disorders) | 3 (3)
Superficial wound dehiscence (Skin and subcutaneous tissue disorders) | 1 (1)
Elective CABG (Cardiac disorders) | 1 (1)
Neck abcess (Infections and infestations) | 1 (1)
Disarthria/TIA (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT01569594/Prot_SAP_000.pdf